CLINICAL TRIAL: NCT03136887
Title: A Prospective, Multicenter, Post-Market Clinical Follow-Up Study to Evaluate the Safety and Effectiveness of the JOURNEY™ II XR Total Knee System
Brief Title: JOURNEY II XR Safety and Effectiveness PMCF
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4049-06; U1111-1191-7751 (Other: WHO)
Record Dates: First submitted 2017-01-25; First posted 2017-05-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Vasculitis With Rheumatoid Arthritis of Knee; Unilateral Post-Traumatic Osteoarthritis of Knee; Knee Osteoarthritis; Degenerative Arthritis Peripheral Joint; Failed Osteotomies; Failed Unicompartmental Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- JOURNEY II XR TKA: This is a single arm study, all subjects will receive JOURNEY II XR TKA
  Interventions: Device: JOURNEY II XR Total Knee System

INTERVENTIONS:
Device: JOURNEY II XR Total Knee System — JOURNEY II XR Total Knee System

SUMMARY:
This study was designed to demonstrate the safety and performance of the JOURNEY II XR total knee system by evaluating implant survival rates at 10 years using Kaplan-Meier analysis. All participants will be implanted with the JOURNEY II XR total knee system.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is considered the most beneficial and cost-effective treatment for end-stage knee arthritis and is the most frequently performed joint replacement surgery. TKA is also indicated for earlier osteoarthritis (OA) interventions, such as osteotomy or unicompartmental replacement, when additional treatment is warranted. One device option available once the decision is made to perform TKA is the JOURNEY II XR Total Knee System. The JOURNEY II XR Total Knee System is designed to be a more "natural feeling" total knee replacement. The goal of the JOURNEY II XR is to enable a higher level of function after total knee replacement by relieving pain and restoring the ability to participate in active lifestyles. The main aim of this study is to generate long-term safety and performance data for the JOURNEY™ II XR Total Knee System. Effectiveness information such as short- and long-term function, subject satisfaction, and quality of life will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. require TKA due to rheumatoid arthritis, post-traumatic arthritis, osteoarthritis, or degenerative arthritis, failed osteotomies, or failed unicompartmental replacement
2. have all cruciate and collateral ligaments intact in the index joint
3. adult patients that in the judgement of the Investigator are skeletally mature
4. be willing and able to participate in required follow-up visits at the investigational site and to complete study procedures and questionnaires
5. consent to participate in the study by signing the IRB/EC approved informed consent form

Exclusion Criteria:

1. have any of the following conditions in the index joint:

   * Intra-articular corticosteroid therapy (or any other intra-articular therapy) in the study knee within 3 months of study enrollment
   * Significant varus or valgus deformities (>15º)
   * Incomplete or insufficient tissue surrounding the knee
   * Collateral ligament insufficiency
   * Inadequate bone stock to support the device (e.g., severe osteopenia/osteoporosis) or will require use of femoral and tibial stems
   * History of prior TKA
2. have any of the following conditions in the contralateral joint:

   * a previous TKA as a revision for a failed total or unicondylar knee arthroplasty
   * a primary TKA or unicondylar knee arthroplasty that is not fully healed and well-functioning as determined by the Investigator
3. have any of the following conditions of the hip:

   * a previous contralateral or ipsilateral revision hip arthroplasty
   * ipsilateral hip arthritis resulting in flexion contracture
   * previously received an ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty that is not fully healed and well-functioning as determined by the Investigator
4. have a diagnosis of an immunosuppressive disorder
5. have an active infection, treated or untreated, systemic or at the site of the planned surgery
6. have conditions that may interfere with the TKA survival or outcome, including but not limited to: Paget's disease, Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, renal insufficiency or neuromuscular disease
7. have a BMI > 40
8. be facing current or impending incarceration
9. have a known allergy to study device or one or more of its components
10. be pregnant or have plans to become pregnant during the course of the study
11. have, in the opinion of the Investigator, an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse
12. be enrolled in another drug, biologic, or device study within 30 days of screening
13. be known to be at risk for lost to follow-up or failure to return for scheduled visits
14. during the surgery, have a cruciate ligament tibial bone island that is secured with any fixative device (e.g. screw, plate, etc.).

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from their orthopedic surgeons practice.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | 10 years
  Did knee survive with no revision through 10 years

SECONDARY OUTCOMES:
Knee function | 10 years
  Lateral Step-Up Test
Quality of Life - EQ-5D - 3L | 10 years
  Patient Reported Outcomes using EuroQol Five Dimensions Questionnaire (EQ-5D - 3L) questionnaire
Quality of Life - FJS | 10 years
  Patient Reported Outcomes using Forgotten Joint Score (FJS) questionnaire
Quality of Life - KOOS | 10 years
  Patient Reported Outcomes using Knee Injury and Osteoarthritic Outcome Scores (KOOS) questionnaire
Quality of Life - ABC scale | 10 years
  Patient Reported Outcomes using Activities-specific Balance Confidence (ABC) questionnaire
Quality of Life - SAPSS | 10 years
  Patient Reported Outcomes using Self-Administered Patient Satisfaction Score (SAPSS) questionnaire
Physiotherapy (PT) utilization - No. of visits | 6 Months Post-operatively
  Number of PT visits required up to 6 months after surgery
Physiotherapy (PT) utilization - Period of visits | 6 Months Post-operatively
  Time period during which PT appointments are required up to 6 months after surgery
Radiographic outcomes | 10 years
  X-rays of index joint
Adverse Events (AEs) | 10 years
  All AEs will be collected and reported

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Loma Linda University Dept. of Orthopaedic Surgery, Loma Linda, California
  - Holy Cross Orthopedic Institute, Fort Lauderdale, Florida
  - Castle Orthopaedics & Sports Medicine, S.C., Aurora, Illinois
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - DeClaire LaMacchia Orthopaedic Institute, Rochester, Michigan
  - Reno Orthopaedic Center, Reno, Nevada
  - Mercer Bucks Orthopaedics, Hamilton, New Jersey
  - NYU Hospital for Joint Diseases / NYU Langone Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Center for Hip & Knee Replacement, New York, New York
  - The Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Providence Regional Medical Center Everett, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh JA, Lewallen DG. Time trends in the characteristics of patients undergoing primary total knee arthroplasty. Arthritis Care Res (Hoboken). 2014 Jun;66(6):897-906. doi: 10.1002/acr.22233. PMID 24249702
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] NIH Consensus Panel. NIH Consensus Statement on total knee replacement December 8-10, 2003. J Bone Joint Surg Am. 2004 Jun;86(6):1328-35. doi: 10.2106/00004623-200406000-00031. No abstract available. PMID 15173310
- [Background] Dowsey MM, Gunn J, Choong PF. Selecting those to refer for joint replacement: who will likely benefit and who will not? Best Pract Res Clin Rheumatol. 2014 Feb;28(1):157-71. doi: 10.1016/j.berh.2014.01.005. PMID 24792950
- [Background] Gidwani S, Fairbank A. The orthopaedic approach to managing osteoarthritis of the knee. BMJ. 2004 Nov 20;329(7476):1220-4. doi: 10.1136/bmj.329.7476.1220. No abstract available. PMID 15550426
- [Background] Parvizi J, Hanssen AD, Spangehl MJ. Total knee arthroplasty following proximal tibial osteotomy: risk factors for failure. J Bone Joint Surg Am. 2004 Mar;86(3):474-9. doi: 10.2106/00004623-200403000-00003. PMID 14996871